CLINICAL TRIAL: NCT01826201
Title: A Phase 2a, Randomized, Blinded, Paired Psoriasis Lesion, Comparative, Placebo-controlled Study to Evaluate the Safety, Preliminary Efficacy and Pharmacokinetics of Epidermal Administrations of MOL4239 in Adults With Plaque Psoriasis
Brief Title: Paired Psoriasis Lesion, Comparative, Study to Evaluate MOL4239 in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moleculin, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M-02
Record Dates: First submitted 2013-03-21; First posted 2013-04-08 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10% MOL4239 ointment & placebo ointment (Experimental): 10% MOL4239 ointment to one target lesion and placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days
  Interventions: Drug: MOL4239; Drug: Placebo

INTERVENTIONS:
Drug: MOL4239 — 10% MOL4239 ointment to one target lesion twice a day for 28.5 consecutive days
Drug: Placebo — placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days

SUMMARY:
The purpose of this study is to determine whether MOL4239 is effective in adult subjects with mild to moderate plaque psoriasis by comparing two target lesions in which each subject will apply MOL4239 ointment to one target lesion and placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days.

DETAILED DESCRIPTION:
This is a phase 2a, Randomized, Multi-center, Blinded, Paired Psoriasis Lesion, Comparative Placebo-Controlled study to evaluate the safety, preliminary efficacy and pharmacokinetics of MOL4239 in 30 adult subjects with mild to moderate plaque psoriasis. Eligible subject will have a diagnosis of mild to moderate plaque psoriasis affecting 9.9% body surface area (BSA) or less, and two designated similar target lesions with a Psoriasis Severity Score of at least 6 or higher. Each subject will apply 10% MOL4239 ointment to one target lesion and placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Adults, males or females, 18 to 72 years of age (both inclusive.)
* Mild to moderate plaque psoriasis with lesions that in total are no more than 9.9% BSA and with a baseline Psoriasis Severity Score (PSS) of 6 or more.
* Identification of bilaterally symmetrical or approximately equivalent target lesions of at least 2.5 x 2.5 cm (~6 cm2) on the trunk, arms or legs to mid calf with a Psoriasis Severity Score (PSS) of 6 or greater.
* Willing to avoid tanning devices or exposure of the treated skin to the sun.
* Willing to not use cosmetics, including lotions, creams, and moisturizers on the treated lesions.
* Use of Eucerin® is allowed on all non-test site areas.
* Willing to forgo systemic and other topical treatments for psoriasis during the course of the study.
* Willing to avoid bathing or swimming for two hours after study drug treatment.
* Negative urine pregnancy test at Screening and baseline for women of childbearing potential (WOCP).
* Sexually active WOCP participating in the study must agree to use a medically acceptable method of contraception while on study.
* Must have recovered from the effects of any surgery, other than minor office surgical procedures, and a minimum of 3 months must have elapsed from the day of surgery to the day of screening.

Exclusion Criteria:

* Presence of significant abnormalities of liver or renal functions.
* Presence of any clinically significant lab abnormalities at screening.
* Any significant uncontrolled medical disease.
* Use of the anti-tumor necrosis factor (TNF) biologic agents 4 months prior to randomization or use of Stelara 6 months prior to randomization.
* Use, within one month prior to baseline or during the study, of: 1) systemic immunosuppressive drugs (e.g., tacrolimus), or 2) oral meds (e.g. methotrexate, retinoids, etc.).
* Use within one month prior to baseline or during the study of: 1) Systemic corticosteroids, 2) Systemic antibiotics, 3) other systemic antipsoriatic treatment, 4) oral psoralen with ultraviolet A (PUVA) therapy, or 5) ultraviolet B (UVB) therapy.
* Use within two weeks prior to baseline or during the study of: 1) topical anti-psoriatic drugs, 2) topical corticosteroids, 3) other topical retinoids, or 4) topical immunosuppressive agents.
* Current diagnosis of unstable forms of psoriasis in the treatment area, including guttate, erythrodermic, exfoliative or pustular psoriasis.
* Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris.
* Females who are pregnant, breast feeding, or planning a pregnancy.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tschen, MD, Principal Investigator — Academic Dermatology Associates; Javier Alonso-Llamazares, MD, Principal Investigator — International Dermatology Research, Inc.; Steven Kempers, MD, Principal Investigator — Minnesota Clinical Study Center
Locations (3):
- United States (3):
  - International Dermatology Research, Inc., Miami, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-site study conducted at three sites in the United States of America. Date first subject enrolled: 22 April 2013 and date last subject completed: 13 August 2013.
Groups:
- 0% and 10% MOL4239 Ointment: 10% MOL4239 ointment to one target lesion and placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days
Period: Overall Study
Arm/Group | 0% and 10% MOL4239 Ointment
Started | 21 (Subjects in each arm are same)
Completed | 17
Not Completed | 4
Not completed — Non compliance with protocol | 4

BASELINE CHARACTERISTICS:
Arm/Group | 10% MOL4239 Ointment & Placebo Ointment
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Day 28 in PSS (Psoriasis Severity Score) of the Treatment Target Lesions Compared to Placebo Target Lesions
Description: he study drug application sites were scored for erythema, induration, and scale assessment using the PSS Scoring system. Psoriasis Severity Score (PSS) Erythema 0 - 4, 0 None, may have residual non-erythematous discoloration
  1 Faint erythema 2 Moderate erythema/red color 3 Severe erythema/very red discoloration 4 Very severe erythema/extreme red coloration Induration 0 - 4 0 None
  1. Trace or slight elevation of plaque above normal skin level
  2. Moderate elevation with rounded or sloped edges to plaque
  3. Marked elevation with hard, sharp edges to plaque
  4. Very marked elevation with very hard, sharp edges to plaque Scaling 0 - 4
  0 None
  1. Fine scales
  2. Coarse scales
  3. Thick scales with a rough surface
  4. Thick scales with a very rough surface
  The scores were summed
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: PSS score
Units Other Than Participants: Target Lesions
Groups:
- 10% MOL4239 Ointment: 10% MOL4239 ointment to one target lesion and placebo ointment to the contralateral target lesion twice a day for 28.5 consecutive days
- Placebo Ointment: 10% MOL4239 to one target lesion and placebo to contralateral target lesion
Arm/Group | 10% MOL4239 Ointment | Placebo Ointment
Number analyzed (Participants) | 17 | 17
Number analyzed (Target Lesions) | 17 | 17
PSS score | -1.9 (1.45) | -1.5 (1.87)

2. Secondary Outcome: Improvement in Lesion Appearance
Description: Photography of the MOL4239 and placebo treated lesions will be performed at baseline, Day 7, Day 14 and Day 28 to assess for the improvement in lesion appearance after drug treatment. The assessment will be completed by a blinded panel of dermatologists experienced in the assessment of psoriasis.
Time Frame: Baseline and Day 28
Reporting Status: Not Posted

3. Secondary Outcome: Physician's Treatment Preference
Description: The physician's treatment preference utilizing visual assessment and selection of the most improved plaque. The determination will be either 1)right lesion is preferred compared to left, 2)left lesion is preferred compared to right, 3) no difference between the right and left lesion.
Time Frame: Day 7, Day 14, Day 28
Population: Per protocol
Measure: Number; unit: participants
Units Other Than Participants: lesions
Arm/Group | 0% and 10% MOL4239 Ointment
Number analyzed (Participants) | 17
Number analyzed (lesions) | 34
participants
  0% ointment treated lesion | 5
  10% ointment treated lesion | 4
  Neither lesion | 8

4. Secondary Outcome: Treatment Success
Description: Percent of patients achieving treatment success in the treatment group compared to the placebo group on day 28. Treatment success is defined as patient achieving a psoriasis severity score (PSS) of 3 or less, or an improvement of 5 points or more on the PSS.
Time Frame: Baseline and Day 28
Reporting Status: Not Posted

5. Secondary Outcome: Change in EIS Area
Description: Change in Erythema, Induration and Scale (EIS) area. Total score will be the EIS x Area, and will be calculated at baseline, Day 7, Day 14 and Day 28. The EIS will represent the sum of individual scores of Erythema, Induration and Scale using the same scale utilized in the PSS. The area of active erythema, induration and scale will be measured and the total scores will be calculated from the EIS scores multiplied by the area in cm2.
Time Frame: Baseline and Day 28
Reporting Status: Not Posted

6. Secondary Outcome: Safety Assessment
Description: Safety will be assessed based on reported adverse events, physical examination, vital signs, electrocardiograms, hematology, serum chemistry and urinalysis. Adverse events will be reported throughout the trial. Vital signs will be performed at screening, baseline, prior to the morning dose on Days 0, 1, 7, 14, 28, and at the follow up visit on Day 42. Physical examinations will be performed at Screening, baseline and Day 28. Hematology, serum chemistry and urinalysis will be performed at screening, baseline, Days 1, 7, 14, 28, and at the follow up visit on Day 42. ECGs will be performed at Screening, baseline and Day 28.
Time Frame: Baseline and Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 0% and 10% MOL4239 Ointment
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0% and 10% MOL4239 Ointment (N=21)
Haematuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor approves content of communication.